CLINICAL TRIAL: NCT03626623
Title: A Prospective, Randomized, Controlled Trial Comparing Cytal Wound Matrix 1-Layer to Standard of Care (SOC) in the Management of Diabetic Foot Ulcers (DFUs)
Brief Title: Diabetic Foot Ulcer Study Comparing Cytal Wound Matrix 1-Layer to Standard of Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor Discretion
Sponsor: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR2017-006
Record Dates: First submitted 2018-06-12; First posted 2018-08-13 (Actual); Results first posted 2021-02-15 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Diabetes; Diabetic Foot; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1
Keywords: Diabetes; Foot Ulcer
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot; Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Foot Ulcer | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard of Care (SOC) (Placebo Comparator): The usual care a licensed health care provider would give patients to treat diabetic foot ulcers or wounds.
  Interventions: Other: Standard of Care (SOC)
- Cytal Wound Matrix 1-Layer (Active Comparator): The application of the Cytal Wound Matrix 1-Layer device according to the Cytal Wound Matrix 1-Layer instructions for use (IFU).
  Interventions: Device: Cytal Wound Matrix 1-Layer

INTERVENTIONS:
Device: Cytal Wound Matrix 1-Layer — Cytal® Wound Matrix 1-Layer is composed of a porcine (pig) derived extracellular matrix known as urinary bladder matrix. It is intended for the management of a variety of wounds.The individual device is intended for one time use.
  Arms: Cytal Wound Matrix 1-Layer
Other: Standard of Care (SOC) — Standard of care (SOC) is defined as the usual care a licensed health care provider would give patients to treat diabetic foot ulcers or wounds. SOC associated procedures and policies may vary across clinical settings.
  Arms: Standard of Care (SOC)

SUMMARY:
This is a two-armed randomized controlled trial (RCT) primarily aimed at determining if application of Cytal Wound Matrix 1-Layer intervention to diabetic foot ulcers shows improved wound closure rates when compared to standard care intervention.

DETAILED DESCRIPTION:
This is a prospective, two-armed, multi-center randomized controlled trial (RCT) comparing Cytal Wound Matrix 1-Layer intervention to standard of care (SOC) intervention in patients presenting with diabetic foot ulcers (DFU). Up to one hundred and fifty patients recruited from US based medical centers and randomized (using a 2(active):1(control) randomization scheme) to receive either Cytal Wound Matrix 1-Layer intervention or standard of care intervention.Complete wound closure incidence, wound healing rates, wound recurrence, and various health related quality of life (HRQOL) outcomes will be compared between study arms. Additionally, a cost effective analysis (i.e. direct and indirect costs) and review of individual and group changes in narcotic prescription patterns will also be evaluated. While incidence of wound closure rates will be evaluated through 12 weeks, protocol defined patient follow-up is for two years.

Data will be captured for remaining study objectives during these two years. An independent biostatistician will review all participant data for power and futility analysis. In addition, a clinical events committee (CEC) will adjudicate all adverse events (AEs) and serious adverse events (SAEs).

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form by subject or legally authorized representative.
2. Stated willingness to comply with all study procedures and availability for the duration of the study. Subject is able and willing to tolerate non-removable offloading device for the duration of the run-in and intervention phases of the study.
3. Subject is male or female and at least 21years of age.
4. Subject has a clinical diagnosis of type 1 or type 2 diabetes.
5. Subject's current foot ulcer(s) has been present for > 30 days and ≤ 365 days.
6. Subject's current foot ulcer(s), post-debridement is/are predominantly below the malleoli and on the plantar surface of the foot.
7. Subject's foot ulcer(s) must be Wagner type 1 or type 2.
8. Post debridement, subject's ulcer(s) are free of necrotic debris and appear to be comprised of healthy, vascularized tissue.
9. All qualifying ulcers are ≥ 5cm away from any other ulcer on the same foot.
10. Subject's ulcer(s) is ≥ 1cm2 and ≤ 20cm2 at randomization (length x width).
11. Subject's HbA1C reading is ≤10%.
12. Subject's Serum Creatinine ≤ 3.0mg/dL.
13. Subject has adequate circulation to the foot as measured by Ankle-Brachial Index (ABI) ≥ 0.7.
14. Negative pregnancy test at randomization for women.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Subject is pregnant, breastfeeding, or unwilling to practice birth control during participation in the study, if applicable.
2. Allergy or hypersensitivity to materials in porcine-based study products (per subject report) or personal preference.
3. Subject report of concurrent participation in another clinical trial that involves a drug.
4. The subject has any condition that, in the Investigator's opinion, would warrant exclusion from the study or prevent the subject from completing the study.
5. Subject has clinical evidence of gangrene on any part of the affected foot.
6. The subject's ulcer(s) is/are due to a non-diabetic etiology, ulcers of arterial, venous stasis, pressure, radiation, traumatic, rheumatoid, vasculitis, collagen vascular disease, or other non-diabetic etiologies.
7. Subject has unstable Charcot foot, Charcot foot with a bony prominence(s) or Charcot amputation.
8. Qualifying wound(s) is connected to another ulcer via a fistula.
9. Subject has one or more medical condition(s) including: renal, hepatic, hematological, neurologic, or immune disease that in the opinion of the Investigator would make the subject an inappropriate candidate for this wound healing study.
10. Subject has or has had a malignant disease (other than basal cell carcinoma) that has not been in remission for at least five years.
11. Subject is receiving oral or parenteral corticosteroids, immunosuppressive or cytotoxic agents, or is anticipated to require such during the course of the study.
12. Subject has acute osteomyelitis of the affected foot.
13. Subject's ulcer(s) is accompanied by active cellulitis.
14. Subject has received growth factor or enzymatic therapy within 2 weeks of consent.
15. Subject is currently receiving or has received radiation, radiologic implants, or chemotherapy.
16. Subject is allergic to any of the primary or secondary dressing materials, including occlusive dressings and the adhesives on such dressings.
17. Subject's ulcer(s) has decreased in size by >30% during the run-in phase.
18. Subject's ulcer(s) has increased in size by >50% during the run-in phase.
19. Subject's ulcer(s) has tunnels or sinus tracts that cannot be completely debrided.
20. Subject has severe malnutrition as evidenced by albumin <2.0 g/dL.
21. Subject has a bleeding disorder as documented by a diagnosis of a bleeding disorder.
22. Subject is on dialysis.
23. Any DFU(s) is infected and has not been treated for any clinically suspected infection prior to application of any product.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2020-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Matthews, Study Chair — Integra LifeSciences
Locations (3):
- United States (3):
  - Limb Preservation Platform, Inc., Fresno, California
  - Louisiana State University Health Science Center (LSUHSC), New Orleans, Louisiana
  - MedStar Health Research Institute, Hyattsville, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen YH, DeMets DL, Lan KK. Increasing the sample size when the unblinded interim result is promising. Stat Med. 2004 Apr 15;23(7):1023-38. doi: 10.1002/sim.1688. PMID 15057876
- [Background] Dumville JC, O'Meara S, Deshpande S, Speak K. Hydrogel dressings for healing diabetic foot ulcers. Cochrane Database Syst Rev. 2013 Jul 12;2013(7):CD009101. doi: 10.1002/14651858.CD009101.pub3. PMID 23846869
- [Background] Wu L, Norman G, Dumville JC, O'Meara S, Bell-Syer SE. Dressings for treating foot ulcers in people with diabetes: an overview of systematic reviews. Cochrane Database Syst Rev. 2015 Jul 14;2015(7):CD010471. doi: 10.1002/14651858.CD010471.pub2. PMID 26171906
- [Background] Bann CM, Fehnel SE, Gagnon DD. Development and validation of the Diabetic Foot Ulcer Scale-short form (DFS-SF). Pharmacoeconomics. 2003;21(17):1277-90. doi: 10.2165/00019053-200321170-00004. PMID 14986739
- [Background] Yazdanpanah L, Nasiri M, Adarvishi S. Literature review on the management of diabetic foot ulcer. World J Diabetes. 2015 Feb 15;6(1):37-53. doi: 10.4239/wjd.v6.i1.37. PMID 25685277
- [Background] Rice JB, Desai U, Cummings AK, Birnbaum HG, Skornicki M, Parsons NB. Burden of diabetic foot ulcers for medicare and private insurers. Diabetes Care. 2014;37(3):651-8. doi: 10.2337/dc13-2176. Epub 2013 Nov 1. PMID 24186882
- [Background] Margolis DJ, Kantor J, Berlin JA. Healing of diabetic neuropathic foot ulcers receiving standard treatment. A meta-analysis. Diabetes Care. 1999 May;22(5):692-5. doi: 10.2337/diacare.22.5.692. PMID 10332667
- See also: Description of Cytal Wound Matrix Products (including Cytal Wound Matrix 1-Layer) — https://acell.com/wound-matrix/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care (SOC) | Cytal Wound Matrix 1-Layer
Started | 5 | 10
Completed | 0 | 0
Not Completed | 5 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SOC) | Cytal Wound Matrix 1-Layer | Total
Number analyzed (Participants) | 5 | 10 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 9 | 14
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 5 | 9 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 10 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Number of Wounds [Number; unit: Wounds] | 5 | 10 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Wounds With Wound Closure
Description: The primary endpoint of the study is to measure the incidence of complete wound closure (defined as 100% epithelialization) between randomized groups. Number of wounds was calculated as the total across all participants.
Time Frame: up to 12 weeks
Population: The study was terminated by sponsor prior to completion, all enrolled subjects did not complete 12 weeks follow-up prior to termination.
Measure: Number; unit: wounds
Arm/Group | Standard of Care (SOC) | Cytal Wound Matrix 1-Layer
Number analyzed (Participants) | 4 | 9
wounds | 1 | 1

2. Secondary Outcome: Wound Size Change
Description: Measure changes in wound size, measured in cm2/week between randomized groups.
Time Frame: up to 12 weeks
Population: The study was terminated by sponsor due to low enrollment and data were not collected.
Arm/Group | Standard of Care (SOC) | Cytal Wound Matrix 1-Layer
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Complete Wound Closure Time
Description: Measure time to complete wound closure between randomized groups.
Time Frame: up to 12 weeks
Population: The study was terminated by sponsor due to low enrollment and data were not collected.
Arm/Group | Standard of Care (SOC) | Cytal Wound Matrix 1-Layer
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Wound Recurrence
Description: Measure wound recurrence after healing is complete between randomized groups.
Time Frame: at 26 week visit and 52 week visit
Population: The study was terminated by sponsor due to low enrollment and data were not collected.
Arm/Group | Standard of Care (SOC) | Cytal Wound Matrix 1-Layer
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Short Form-20 (SF-20)
Description: The Short Form-20 is a 20-item questionnaire used to assess generic health outcomes from the participant's perspective. Scores are linearly measured from 0 (worst) to 100 (best) health functioning scores, respectively.
Time Frame: Baseline visit, visit #7, visit #13, 26 wk. visit, and 52 wk.visit
Population: The study was terminated by sponsor due to low enrollment and data were not collected.
Arm/Group | Standard of Care (SOC) | Cytal Wound Matrix 1-Layer
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Diabetic Foot Ulcer Scale- Short Form (DFS-SF)
Description: The diabetic foot ulcer scale- short form (DFS-SF) is a 29-item questionnaire designed to assess the impact of diabetic foot ulcers (DFUs) and their intervention on quality of life of participants diagnosed with diabetes. Scores measured from 0 (lower) to 100 (higher) quality of life, respectively.
Time Frame: Baseline visit, 26 week visit, and 52 week visit
Population: The study was terminated by sponsor due to low enrollment and data were not collected.
Arm/Group | Standard of Care (SOC) | Cytal Wound Matrix 1-Layer
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Visual Analogue Scale (VAS) for Pain
Description: The visual analogue scale (VAS) is a psychometric response scale for pain. It measures subjective characteristics or attitudes regarding perceived pain levels from participants. Participants are asked to draw a vertical line on a 10 cm horizontal line indicating what their current pain level would be. The distance between the start of the horizontal line to the vertical line is calculated in cm with a higher score (100) indicating greater pain intensity.
Time Frame: Up to 52 week visit (until study completion)
Population: The study was terminated by sponsor due to low enrollment and data were not collected.
Arm/Group | Standard of Care (SOC) | Cytal Wound Matrix 1-Layer
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Katz Index of Independence in Activities of Daily Living (KATZ ADL)
Description: The Katz ADL is a 6-item questionnaire measuring independence in activities of daily living such as bathing, dressing, toileting, transfers, feeding, and continence. Each item is dichotomized as either having a score of zero (i.e. dependence) or one (i.e. independence). This will be completed with the aid of a trained study staff member.
Time Frame: Baseline visit, visit 7, visit 13, 26 wk visit, and 52 wk visit
Population: The study was terminated by sponsor due to low enrollment and data were not collected.
Arm/Group | Standard of Care (SOC) | Cytal Wound Matrix 1-Layer
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Adverse Events Frequency
Description: This outcome measures diabetic foot ulcer (DFU) related adverse event frequency including unexpected adverse device events (UADEs) or serious adverse experiences (SAEs) throughout the duration of the study as well as evaluate such adverse event frequencies between randomized groups.
Time Frame: up to 52 week visit (until study completion)
Population: The study was terminated by sponsor due to low enrollment and data were not collected.
Arm/Group | Standard of Care (SOC) | Cytal Wound Matrix 1-Layer
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Narcotic Prescription Changes Between Trial Arms
Description: This outcome measures changes in number of diabetic foot ulcer (DFU) related narcotic prescriptions by study participant and between randomized groups.
Time Frame: up to 52 week visit (until study completion)
Population: The study was terminated by sponsor due to low enrollment and data were not collected.
Arm/Group | Standard of Care (SOC) | Cytal Wound Matrix 1-Layer
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Participant Ambulatory Status
Description: This outcome measures any changes in ambulatory status (i.e. bed, wheel chair, walk w/ assistance, or walk independent) by study participant and between randomized groups.
Time Frame: up to 52 week visit (until study completion)
Population: The study was terminated by sponsor due to low enrollment and data were not collected.
Arm/Group | Standard of Care (SOC) | Cytal Wound Matrix 1-Layer
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Return to Work Status
Description: This outcome measures differences in "return to work status" and/or "reported work status", activities of daily living, or disability status by study participant and between randomized groups.
Time Frame: up to 52 week visit (until study completion)
Population: The study was terminated by sponsor due to low enrollment and data were not collected.
Arm/Group | Standard of Care (SOC) | Cytal Wound Matrix 1-Layer
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Diabetic Foot Ulcer (DFU) Specific Ancillary Medical Care
Description: This outcome measures the incidence of diabetic foot ulcer (DFU) specific related medical care a study participant receives outside of the medical care provided by the investigator. Examples of ancillary care include, but are not limited to, emergency room (ER) visits, urgent care visits, outside medical procedures such as surgery, etc. The incidence of subjects requiring ancillary medical care will be tabulated and compared between randomized groups. This data will be collected via two questions (i.e. "Did participant receive any ancillary medical care?" and "If "yes", then specify where"). Responses are verified using source documentation.
Time Frame: up to 52 week visit (until study completion)
Population: The study was terminated by sponsor due to low enrollment and data were not collected.
Arm/Group | Standard of Care (SOC) | Cytal Wound Matrix 1-Layer
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Diabetic Foot Ulcer (DFU) Related Direct Product(s) Costs
Description: This outcome measures direct costs of the products by total cost per subject stratified by healed vs. non healed DFU.
Time Frame: up to 52 week visit (until study completion)
Population: The study was terminated by sponsor due to low enrollment and data were not collected.
Arm/Group | Standard of Care (SOC) | Cytal Wound Matrix 1-Layer
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Indirect Diabetic Foot Ulcer (DFU) Product(s) Costs
Description: This outcome measures total indirect and incidental costs of diabetic foot ulcer products used per study participant by each visit.
Time Frame: up to 52 week visit (until study completion)
Population: The study was terminated by sponsor due to low enrollment and data were not collected.
Arm/Group | Standard of Care (SOC) | Cytal Wound Matrix 1-Layer
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 weeks
Arm/Group | Standard of Care (SOC) | Cytal Wound Matrix 1-Layer
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/5 | 3/10
Other Adverse Events (participants affected / at risk) | 3/5 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SOC) (N=5) | Cytal Wound Matrix 1-Layer (N=10)
chest pain (Cardiac disorders) | 0 (0) | 1 (1)
infection of target wound/ulcer (Infections and infestations) | 0 (0) | 2 (2)
cellulitis of target wound/ulcer (Infections and infestations) | 2 (2) | 0 (0)
elbow infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SOC) (N=5) | Cytal Wound Matrix 1-Layer (N=10)
flash burn, eye (Eye disorders) | 0 (0) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
common cold (General disorders) | 0 (0) | 1 (1)
wound recurrence (after closure) (General disorders) | 0 (0) | 1 (1)
new toe wound on target foot (General disorders) | 1 (1) | 1 (1)
new wound on non-target limb (General disorders) | 0 (0) | 1 (1)
thumb infection (Infections and infestations) | 1 (1) | 0 (0)
cellulitis, leg (Infections and infestations) | 1 (1) | 1 (1)
infection of target wound (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to early termination, additional primary and secondary endpoint analyses were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT03626623/Prot_SAP_000.pdf